CLINICAL TRIAL: NCT02722681
Title: Developing a Biomarker for Monitoring Clinical Outcomes in Children With Spinal Lipoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Institute of Child Health (Other)
Collaborators: Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 13ND18
Record Dates: First submitted 2016-03-16; First posted 2016-03-30 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2016-03

CONDITIONS: Lipoma of Spinal Cord
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be stored during length of project.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Symptomatic spinal lipoma patients: Spinal lipoma patients undergoing surgery due to symptomatic lipoma. Routine blood and urine samples will be taken pre-operatively, some will be kept aside for research. Cerebrospinal fluid is drained intraoperatively and usually discarded, some will be kept for research.
  Interventions: Procedure: Blood and urine sampling; Procedure: Cerebrospinal fluid sampling
- Asymptomatic spinal lipoma patients: Spinal lipoma patients who remain asymptomatic. Routine blood and urine samples will be taken as part of routine clinical care, some will be kept for research.
  Interventions: Procedure: Blood and urine sampling
- Non-lipoma spinal conditions: Patients undergoing spinal surgery for a non-lipoma related condition. Routine blood and urine samples will be taken pre-operatively, some will be kept aside for research. Cerebrospinal fluid is drained intra-operatively and usually discarded, some will be kept for research.
  Interventions: Procedure: Blood and urine sampling; Procedure: Cerebrospinal fluid sampling

INTERVENTIONS:
Procedure: Blood and urine sampling — Collection of blood and urine samples taken during usual clinical management
Procedure: Cerebrospinal fluid sampling — Collection of cerebrospinal fluid samples taken during usual clinical management
  Groups: Non-lipoma spinal conditions; Symptomatic spinal lipoma patients

SUMMARY:
'Spinal lipoma' is a condition, present from before birth, in which fatty tissue (lipoma) is attached to the lower end of the spinal cord, tethering it within the vertebral canal. The cord normally moves up and down with respiration, whereas tethering prevents this movement, and can lead to progressive neurological deterioration. The cord and spinal nerves become stretched and their blood supply is damaged irreversibly. Disability may include weakness or pain in the lower body, and urinary disorders in young children. Treatment is surgical, to remove the lipoma and mobilise the spinal cord, with 60 such operations performed per year at Great Ormond Street Hospital. This project aims to develop lipidomic biomarkers in order to predict which children with spinal lipoma are at highest risk of neurological deterioration, and require early surgery, while providing evidence to adopt a more conservative approach for those at lower risk.

DETAILED DESCRIPTION:
Clinical study to seek a metabolic biomarker(s), detectable by mass spectrometry, that can be used to 'stratify' patients with asymptomatic lipoma. In view of the often extensive nature of lipomas associated with the low spinal cord, we hypothesise that lipid components, or metabolites derived from them, may gain entry to the child's bloodstream. The more infiltrative lipomas carry a higher risk of symptomatic deterioration and, we argue, should also have a higher chance of generating a lipid 'signature' in the blood and/or urine. Phase 1 - Cerebrospinal fluid, blood and urine samples will be obtained from patients with spinal lipoma undergoing surgery (n = 3 to 5). Informed consent, following appropriate ethics committee approval, will be implemented. Blood and urine will be sampled pre-operatively, and intra-operative cerebrospinal fluid samples will be obtained. Mass spectrometry analysis will identify lipid species present in the cerebrospinal fluid of these patients, and the extent to which these are also detectable in the patient's blood and/or urine. Any lipid species detected in both cerebrospinal fluid and blood/urine will represent potential biomarkers, and will form the focus of the next phase of the study. Phase 2 will then assess the discriminatory value of these potential biomarkers by comparing their profiles in blood and/or urine from three clinical groups: (i) Patients with spinal lipomas who have neurological symptoms/signs, and are attending hospital for surgery (i.e. similar patients as in Phase 1). Blood/urine samples will be taken preoperatively, to represent the 'high risk' group. (ii) Patients with spinal lipomas who have remained asymptomatic after several years follow-up.

These represent the 'low risk' group; (iii) Patients with spinal conditions not involving lipoma. These represent our 'negative' control group. Group sizes will be determined by power calculations using variance data from the patient measurements in Phase 1. Statistical analysis will be by 1-way ANOVA, or non-parametric equivalent, to test for significant differences between the three groups. Mass spectrometry (Figure 2) will be performed in the Institute of Child Health Centre for Proteomics, Metabolomics and Lipidomics using nano ultra performance liquid chromatography and ultra performance convergence chromatography - quadrupole time of flight mass spectrometry, a new mass spectral technology for lipidomic and metabolomic analysis. Ultra performance convergence chromatography is a chromatography technology that uses carbon dioxide present in a super critical fluid state as a mobile phase and allows the fractionation of metabolites and lipids according to their class and not hydrophobicity. It enables quantitation of all the major lipid classes present in a tissue including phospholipids, free fatty acids, esterified fatty acids, cholesterol esters and sterols. Non-lipid molecules (e.g. choline) might also show altered abundance in lipoma patients and so a more general metabolomics analysis will also be undertaken, if time permits.

ELIGIBILITY:
Inclusion Criteria:

* patient with proven spinal lipoma

Exclusion Criteria:

* complex spinal lipomas related to other developmental abnormalities

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children under the age of 16 attending GOSH for management of spinal lipomas and non-lipoma related spinal conditions
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2016-02; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Lipid signature within blood or urine samples of patients with symptomatic spinal lipomas | 2 years
  Lipid profiles from urine and blood samples from spinal lipoma patients will show specific lipids present at a higher concentration in symptomatic patients when compared with asymptomatic patients.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Copp, PhD, Study Chair — Institute of Child Health, UCL; Dominic Thompson, FRCS, Study Director — Great Ormond Street Hospital NHS Trust; Kevin Mills, PhD, Study Director — Institute of Child Health, UCL
Locations (1):
- Institute of Child Health, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No